CLINICAL TRIAL: NCT00556010
Title: Intraoperative Three Dimensional Fluoroscopy Compared to Standard Fluoroscopy for the Assessment of Reduction of Ankle Fractures With Syndesmosis Disruption
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: WEIL-HMO-CTIL
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2011-04

CONDITIONS: Ankle Injuries
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Ankle fractures are common injuries that are being operated routinely. In order to restore the long term function and prevent arthritis of the ankle the broken fragments should be put in place precisely. Inadequate reduction can result in pain and long term disability. Recently, based on MRI studies and clinical studies, a significant number of ankle fractures are apparently fixed with less than optimal results. We suggest that the use of a new device that enables better three dimensional imaging will improve the quality of operations performed for ankle fractures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unstable ankle fractures (as classified by the AO as 44B 44C by Lauge Hansen PER4 or SER4) amenable to open reduction and internal fixation.
2. Patients with syndesmotic rupture as evident from the injury films or during clinical testing in the OR be included in the study.
3. Intraoperative testing will include both a cotton Test and a stress view obtained after bimalleolar fixation has been attained.
4. A positive syndesmotic injury will be defined by the criteria of Pettrone et al as follows: a tib/fib clear space >5mm or tib/fib overlap of <10mm (on the AP view), or a tib/fib overlap of <1mm on the mortise view.

Exclusion Criteria:

1. Patients with a pilon fracture (i.e. plafond fractures AO type 43B and C) will be excluded even if associated with a fibula fracture and syndesmosis disruption.
2. Patients with contraindications to operative treatment and diabetics
3. Women of childbearing age will be excluded if they present with a positive pre-op Beta HCG test or if they refuse a B HCG test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with fracture in the ankle with Syndesmosis disruption
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yorm A Weil, M.D, Principal Investigator — Hadassah Medical Organization; Roy Davidovitch, MD, Study Chair — NYU school of Medicine, Hospital for Joint Diseases , New York, U.S.A; Rami Mosheiff, MD, Study Chair — Hadassah Medical Organization; Kenneth Egol, M.D, Study Chair — NYU school of Medicine, Hospital for Joint Diseases, New York, USA; Amal Khoury, MD, Study Chair — Hadassah Medical Organization; Meir Liebergall, MD, Study Director — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization., Jerusalem, Israel

REFERENCES:
- [Derived] Davidovitch RI, Weil Y, Karia R, Forman J, Looze C, Liebergall M, Egol K. Intraoperative syndesmotic reduction: three-dimensional versus standard fluoroscopic imaging. J Bone Joint Surg Am. 2013 Oct 16;95(20):1838-43. doi: 10.2106/JBJS.L.00382. PMID 24132357